CLINICAL TRIAL: NCT03198130
Title: An Exploratory Tumor Biopsy-Driven Study to Understand the Relationship Between Biomarkers and Clinical Response in Immunomodulatory Treatment-Naïve Patients With Recurrent and/or Metastatic Squamous Cell Carcinoma of Head and Neck Receiving REGN2810 (Anti-PD-1)
Brief Title: An Exploratory Tumor Biopsy-driven Study to Understand the Relationship Between Biomarkers and Clinical Response in Patients With Head and Neck Cancer Receiving REGN2810 (Anti-PD-1)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R2810-ONC-1655; 2016-004029-18 (EudraCT Number)
Record Dates: First submitted 2017-06-19; First posted 2017-06-23 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Recurrent Squamous Cell Carcinoma of Head; Recurrent Squamous Cell Carcinoma of Neck; Metastatic Squamous Cell Carcinoma of Head; Metastatic Squamous Cell Carcinoma Neck
MeSH Terms: interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- REGN2810 (Experimental): REGN2810 administered IV over a 30 minute infusion
  Interventions: Drug: REGN2810

INTERVENTIONS:
Drug: REGN2810 — Intravenous (IV) use
  Other Names: cemiplimab; Libtayo

SUMMARY:
This study is being conducted to compare the relationship of patient response to treatment to changes in tumor microenvironment.

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologically confirmed diagnosis of recurrent and/or metastatic SCCHN (squamous cell carcinoma of the head and neck) with no curative options with at least 1 lesion that is measurable by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria and accessible for biopsies. Primary tumor sites of oral cavity, oropharynx, larynx, or hypopharynx are included.
2. Have failed/are refractory to at least first line chemotherapy OR deemed unsuitable candidate for first line chemotherapy due to medical co-morbidities or patient preference
3. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
4. Adequate hepatic function
5. Adequate renal function
6. Adequate bone marrow function
7. Provide signed informed consent
8. Willing and able to comply with clinic visits and study-related procedures

Key Exclusion Criteria:

1. Ongoing or recent (within 5 years) evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments, which may suggest risk for immune-related adverse event (irAEs)
2. Prior treatment with an agent that blocks the programmed death-1/programmed death-ligand 1 (PD-1/PD-L1) pathway
3. Prior treatment with other immune modulating anti-cancer agents
4. Untreated or active brain metastases or spinal cord compression
5. Immunosuppressive corticosteroid doses within 4 weeks prior to the first dose of REGN2810
6. Prior treatment with idelalisib

Other protocol-defined inclusion/exclusion criteria will apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2020-02-21 (Actual)

PRIMARY OUTCOMES:
Correlation between changes in the tumor microenvironment and the change in tumor volume following REGN2810 treatment versus baseline. | At baseline and during REGN2810 treatment up to week 24

SECONDARY OUTCOMES:
Correlation between baseline tumor characteristics and the change in tumor volume following REGN2810 treatment | At baseline and during REGN2810 treatment up to week 24
Number of participants with treatment-related adverse events | Up to 54 weeks
Concentrations of REGN2810 in serum | Up to 54 weeks
Anti-REGN2810 antibody levels | Up to 54 weeks
The overall response rate (ORR) in patients treated with REGN2810 | Up to 54 weeks
The progression-free survival (PFS) in patients treated with REGN2810 | Up to 54 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (6):
- South Korea (3):
  - Seoul National University, Seoul
  - Yonsei University College of Medicine, Severence Hospital, Seoul
  - Samsung Medical Center, Seoul
- United Kingdom (3):
  - University Birmingham, Birmingham
  - Guy's and St. Thomas' NHS Foundation Trust, London
  - Royal Cancer Hospital, London